CLINICAL TRIAL: NCT03171662
Title: Imaging and Histopathological Examination for Evaluation of Pediatric Appendicitis Score ( PAS ) as a Diagnostic Tool for Acute Appendicitis in Children
Brief Title: Imaging and Histopathological Examination for Evaluation of Pediatric Appendicitis Score
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Michael Samir Rateeb, principle investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PASE
Record Dates: First submitted 2017-05-27; First posted 2017-05-31 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Appendicitis Acute
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group study (Experimental): Imaging and Histopathological examination for Evaluation of Pediatric Appendicitis Score
  Interventions: Other: Evaluation of Pediatric Appendicitis Score

INTERVENTIONS:
Other: Evaluation of Pediatric Appendicitis Score — Imaging and Histopathological examination for Evaluation of Pediatric Appendicitis Score

SUMMARY:
Appendicitis is the most common abdominal disease requiring surgery in children. The risk of developing appendicitis during a lifetime is reported to be 8.7% for boys and 6.7% for girls. Despite its high incidence, there are still diagnostic difficulties. The overall negative appendectomy rate among all children is suggested to be 8.4%, but in children under 6 years of age, the rate has been reported to be as high as 56.7% . The diagnosis of acute appendicitis is considered to be especially challenging in children due to difficulties in communication and examination.

DETAILED DESCRIPTION:
The diagnostic difficulties result in increased risks of both negative appendectomies and a delayed diagnosis, both leading to increased morbidity, more complications, longer hospital stay, and higher costs. These risks are further increased in the younger children. The doctor delay is a known cause contributing to late diagnosis in young children. Other studies, with patients under 3 years and 4 years of age, have found parent delay to contribute as well to the late diagnosis. Our clinical experience, confirmed by the literature, shows that the younger children with acute appendicitis deviate from the typical presentation and clinical findings observed in older children with acute appendicitis.

The use of a clinical score, based on patient history and examination, is one way to possibly improve the diagnostic procedure. There are several available scores. In this systematic review, Pediatric Appendicitis Score (PAS) were considered the most reliable. Pediatric Appendicitis Score is the only score specifically developed for children, composed by Samuel in 2002 when analyzing children between 4 and 15 years of age. Pediatric Appendicitis Score has been validated and recommended by some authors, but only one of these studies has included children less than 4 years of age.

We hypothesized that PAS could be helpful in diagnosing young children with appendicitis and that we would find both parent delay and doctor delay contributing to the often late diagnosis in this age group. The aims of this study were to (1) evaluate Pediatric Appendicitis Score in children, operated on for suspected appendicitis, with respect to Pediatric Appendicitis Score sensitivity, specificity, positive predictive value, and negative predictive value; (2) investigate if there was a delay in diagnosing appendicitis; and (3) identify factors responsible for the possible late diagnosis in younger children In order to improve the diagnostic accuracy of acute appendicitis, ultrasound, computed tomography and post-appendectomy histopathological examination have been used as clinical aids in cutting down the rate of negative appendectomy without increasing morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Children (1-15 years old) coming to hospital with abdominal pain and diagnosed provisionally as acute appendicitis .

Exclusion Criteria:

1. Children below 1 year old or above 15 years old.
2. Complicated appendicitis ( mass or abcess ).
3. Patient with recent history of any abdominal surgeries.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
pediatric appendicitis score | 2 days
  post-appendectomy histopathology

IPD SHARING:
Plan to Share IPD: No